CLINICAL TRIAL: NCT01456936
Title: A Phase 4, Randomized, Double-blind, Active And Placebo-controlled, Multicenter Study Evaluating The Neuropsychiatric Safety And Efficacy Of 12 Weeks Varenicline Tartrate 1mg Bid And Bupropion Hydrochloride 150mg Bid For Smoking Cessation In Subjects With And Without A History Of Psychiatric Disorders
Brief Title: Study Evaluating The Safety And Efficacy Of Varenicline and Bupropion For Smoking Cessation In Subjects With And Without A History Of Psychiatric Disorders
Acronym: EAGLES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051123; 2010-022914-15 (EudraCT Number); EAGLES (Other: Alias Study Number)
Record Dates: First submitted 2011-10-14; First posted 2011-10-21 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; psychiatric disease
MeSH Terms: conditions — Smoking Cessation; Mental Disorders | interventions — Varenicline; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- placebo (Placebo Comparator): Subjects randomized to placebo will receive placebo treatments for all three study drugs. Blinded placebo will be provided for varenicline, bupropion hydrochloride and transdermal nicotine patch (NRT). In addition, subjects will receive blinded placebo treatments for the study drugs they are not randomized to receive.
  Interventions: Drug: Placebo
- varenicline (Active Comparator)
  Interventions: Drug: varenicline tartrate
- bupropion (Active Comparator)
  Interventions: Drug: bupropion hydrochloride
- Nicotine Replacement Therapy Patch (Active Comparator)
  Interventions: Drug: Nicotine Replacement Therapy Patch

INTERVENTIONS:
Drug: Placebo — Triple dummy placebo for each treatment arm
  Arms: placebo
Drug: varenicline tartrate — Subjects will be titrated to the full dose during the first week in the following manner: 0.5 mg (tablet form) once a day for 3 days, 0.5 mg twice a day for 4 days, then 1 mg twice a day for 11 weeks
  Other Names: Chantix; Champix
  Arms: varenicline
Drug: bupropion hydrochloride — Subjects will receive 150 mg (tablet form) once a day for 3 days and then will take 150 mg twice a day for the remainder of the treatment period (11 weeks and 4 days).
  Arms: bupropion
Drug: Nicotine Replacement Therapy Patch — Subjects will start active dosing the morning of the Week 1 visit and will receive a 21 mg transdermal patch per day x 7 weeks, followed by a 14 mg transdermal patch per day x 2 weeks, and then a 7 mg transdermal patch x 2 weeks for a total of 11 weeks of treatment.
  Other Names: NRT
  Arms: Nicotine Replacement Therapy Patch

SUMMARY:
This study is being conducted to assess varenicline and bupropion as aids to smoking cessation treatment in subjects with and without an established diagnosis of major psychiatric disorder and to characterize the neuropsychiatric safety profile (pre-specified adverse events (AEs) in both of these populations).

ELIGIBILITY:
Inclusion Criteria:

* Male or female cigarette smokers, 18- 75 years, motivated to stop smoking and considered suitable for a smoking cessation attempt.
* Smoked an average of at least 10 cigarettes per day during past year and during the month prior to the screening visit, and exhaled carbon monoxide (CO) >10 ppm at screening.
* For Neuropsychiatric cohort- subjects must have proper diagnosis as outlined in protocol.

Exclusion Criteria:

* Subjects with a past or current diagnosis of one of the following disorders:

  a. Psychotic Disorders:
* Schizophreniform
* Delusional Disorder
* Psychotic Disorder NOS b. All Delirium, Dementia, and Amnestic and Other Cognitive Disorders c. All Substance Induced Disorders (Other than nicotine)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8144 (Actual)
Dates: Start 2011-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (156):
- United States (77):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - NoesisPharma Research, Phoenix, Arizona
  - Pharmacology Research Institute, Encino, California
  - Synergy Clinical Research of Escondido, Escondido, California
  - Sun Valley Research Center, Imperial, California
  - Omega Clinical Trials, La Habra, California
  - Pacific Treatment and Research Center UC San Diego Health System, La Jolla, California
  - Pharmacology Research Institute, Los Alamitos, California
  - David Geffen School of Medicine at University of California, Los Angeles, Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - North County Clinical Research, Oceanside, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - University of Colorado Denver, Anschutz Medical Campus , Behavioral Health and Wellness Program, Aurora, Colorado
  - Western Affiliated Research Institute, Denver, Colorado
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Broward Research Group, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Clinical Neuroscience Solutions,Inc., Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - Renstar Medical Research, Ocala, Florida
  - Ocala Psychiatric Associates, Ocala, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Meridien Research, Tampa, Florida
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Northwest Neurobehavioral Health, Meridian, Idaho
  - AMR-Baber Research Inc., Naperville, Illinois
  - American Health Network of IN, LLC, Indianaopolis, Indiana
  - Davis Clinic, Incorporated, Indianapolis, Indiana
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Kentucky Research Group, Louisville, Kentucky
  - A Professional Corporation dba The Center for Sexual Health, Metairie, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Community Clinical Services, Lewiston, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Milford Emergency Associates, Incorporated, Milford, Massachusetts
  - Rahim Shafa, MD, Milford, Massachusetts
  - University of Minnesota- TC, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - The Center for Pharmaceutical Research, PC, Kansas City, Missouri
  - Mercy Health Research, St Louis, Missouri
  - University of Medicine and Dentistry of New Jersey-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Global Medical Institutes LLC; Princeton Medical Institute Woodlands Professional Building, Princeton, New Jersey
  - Social Psychiatry Research Institute Clinical Trials LLC, Brooklyn, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Tooley Group, Cary, North Carolina
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - Wake Internal Medicine Consultants, Inc, Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Southeastern PA Medical Institute, Broomall, Pennsylvania
  - Belmont Center for Comprehensive Treatment, Philadelphia, Pennsylvania
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - East Side Clinical Laboratory, Lincoln, Rhode Island
  - Lincoln Research, Lincoln, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Clinical NeuroScience Solutions, Inc., Memphis, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - James G. Kyser, MD, Nashville, Tennessee
  - FutureSearch Clinical Trials, L.P., Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Peninsula Psychotherapy Center, LLC, Newport News, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Argentina (2):
  - Centro Medico Dra. De Salvo, Ciudad Autonoma de Bs. As, Buenos Aires
  - Centro de Investigacion Clinica WM, Mataderos, Buenos Aires
- Australia (2):
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Monash Alfred Psychiatry Research Centre, Melbourne, Victoria
- Brazil (5):
  - Hospital de Messejana Dr. Carlos Alberto Studart Gomes, Fortaleza, Ceará
  - Irmandade da Santa Casa de Misericórdia Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS - Uniao Brasileira de Educacao e Assistencia, Porto Alegre, Rio Grande do Sul
  - Hospital e Maternidade Celso Pierro - Pontifícia Universidade Católica de Campinas - Campus II, Campinas, São Paulo
  - Instituto Jaqueline Scholz Issa e Mario Issa de cardiologia S/C Ltda, São Paulo, São Paulo
- Bulgaria (10):
  - Mental Health Center "Prof. Dr. Ivan Temkov-Bourgas" Ltd., Burgas
  - MBAL Dr. Hristo Stambolski EOOD, Kazanlak
  - DPB Sv. Ivan Rilski, Novi Iskar
  - UMBAL Dr. Georgi Stranski EAD,, Pleven
  - UMBAL Sveti Georgi EAD, Klinika po psihiatriya, Plovdiv
  - SBALPFZ - Ruse EOOD, Rousse
  - Tsentar za psihichno zdrave - Ruse EOOD, Rousse
  - Meditsinski Tsentar ¿Sveti Naum¿ EOOD, Sofia
  - MHATNP Sveti Naum SJsc., Sofia
  - Specializirana Bolnitsa za Aktivno Lechenie na Belodrobni Bolesti-Troyan EOOD,, Troyan Municipality
- Canada (8):
  - Hamilton Medical Research Group, Hamilton, Ontario
  - Medical Research Associates, Mississauga, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Dr. Felix Yaroshevsky, Toronto, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
  - Centre of Addiction and Mental Health Pharmacy, Toronto, Ontario
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Chile (2):
  - Hospital Regional de Talca, Unidad de Enfermedades Respiratorias, Talca, Maule Region
  - Centro Respiratorio Integral (CENRESIN Ltda.), Quillota, Valparaiso, V Region
- Denmark (2):
  - CCBR A/S, Ballerup Municipality
  - CCBR A/S, Vejle
- Finland (6):
  - Mehiläinen Leppävaara, Espoo
  - Savon Psykiatripalvelu Oy, Kuopio
  - Mehiläinen Nummela, Nummela
  - Oulu Mentalcare, Oulu
  - Porin Lääkäritalo Oy, Pori
  - PEL, Psykiatrian ErikoiLääkärit, Turku
- Germany (7):
  - Klinische Forschung Hamburg GmbH, Hamburg, Hamburg
  - ZSL - Zentrum fuer Medizinische Studien Leipzig GmbH, Leipzig, Saxony
  - Klinische Forschung Berlin-Mitte GmbH, Berlin, State of Berlin
  - emovis GmbH, Berlin, State of Berlin
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Ludwig Maximilians-Universitaet Muenchen, München
  - Universitaetsklinik Tuebingen, Tübingen
- Mexico (4):
  - Centro Respiratorio de Mexico S.C., México, D.f.
  - Consultarios de Medicina Especializada del Sector Privado, Colonia Hipodromo Condesa, Mexico DF
  - Clinica de Enfermedades Cronicas y de Procedimientos Especiales S.C., Morelia, Michoacán
  - Centro de Estudios Clinicos y Especialidades Medicas S.C., Monterrey, Nuevo León
- Lakeland Clinical Trials, Rotorua, New Zealand
- Russia (10):
  - FSBI "Federal Medical Research Center of Psychiatry and Addiction Medicine", Moscow
  - FSBI Moscow Scientific Research Institute of Psychiatry", Moscow
  - Moscow State Public Healthcare Institution Mental Clinical Hospital #1 n.a. N.A. Alexeeva, Moscow
  - Clinical Mental Hospital #12 of Moscow Healthcare Department, Moscow
  - Clinical Psychiatric Hospital #1 of Nizhni Novgorod, Nizhny Novgorod
  - St. Petersburg State Healthcare Institution, St. Nikolay Chudotvorets Mental Hospital, Saint Petersburg
  - FSBI "Saint-Petersburg Scientific Research Psychoneurological Institute n.a. V.M. Bekhterev" of MoH, Saint Petersburg
  - State Healthcare Institution "Psychoneurological Dispensary #2, Saint Petersburg
  - SBEI HPE ##Smolensk State Medical Academy## of MoH of RF, Smolensk
  - Smolensk State Medical Academy of Ministry of Healthcare of Russian Federation, Smolensk
- Slovakia (5):
  - Psychiatricka ambulancia, Mentum, s.r.o., Bratislava
  - Vavrusová consulting s.r.o., Nestatna psychiatricka ambulancia, MUDr. Livia Vavrusova, PhD, Bratislava
  - Psychiatricka ambulancia MUDr. Nada Kuriackova, s.r.o., Levice
  - Psychiatricka ambulancia, PsychoLine s.r.o., Rimavská Sobota
  - Nemocnica s poliklinikou sv. Barbory Roznava a.s., Rožňava
- South Africa (9):
  - Flexivest Fourteen Research Center, Bellville, Cape Town
  - Worthwhile Clinical Trials, Benoni, Johannesburg, Gauteng
  - Vista Clinic, Centurion, Gauteng
  - Soweto Clinical Trials Centre, Johannesburg, Gauteng
  - I Engelbrecht Research Pty, Ltd, Lyttelton, Gauteng
  - Midrand Medical Centre, Midrand, Gauteng
  - Private Practice, Durban, KwaZulu-Natal
  - Randles Road Medical Centre, Durban, KwaZulu-Natal
  - Dr John OBrien Incorporated, Cape Town, Western Cape
- Spain (6):
  - Hospital de La Santa Creu I Sant Pau, Barcelona, Barcelona
  - Hospital General Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic I Provincial, Barcelona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres, Caceres
  - Unidad Especializada en Tabaquismo de la Comunidad de Madrid, Madrid, Madrid
  - Centro de Salud Torrero La Paz, Zaragoza, Zaragoza

REFERENCES:
- [Derived] Daniel B, Lawrence DE, McKenna BS, Saccone P, McRae T, Evins AE, Anthenelli RM. Do tobacco regulatory and economic factors influence smoking cessation outcomes? A post-hoc analysis of the multinational EAGLES randomised controlled trial. BMJ Open. 2024 Sep 20;14(9):e079092. doi: 10.1136/bmjopen-2023-079092. PMID 39306350
- [Derived] Tonnesen P, Lawrence D, Tonstad S. Medication-assisted quit rates in participants with smoking-related diseases in EAGLES: Post hoc analyses of a double-blind, randomized, placebo-controlled clinical trial. Tob Induc Dis. 2022 May 10;20:46. doi: 10.18332/tid/146567. eCollection 2022. PMID 35611069
- [Derived] Cinciripini PM, Kypriotakis G, Green C, Lawrence D, Anthenelli RM, Minnix J, Blalock JA, Beneventi D, Morris C, Karam-Hage M. The effects of varenicline, bupropion, nicotine patch, and placebo on smoking cessation among smokers with major depression: A randomized clinical trial. Depress Anxiety. 2022 May;39(5):429-440. doi: 10.1002/da.23259. PMID 35535436
- [Derived] Ebbert JO, Jimenez-Ruiz C, Dutro MP, Fisher M, Li J, Hays JT. In Reply: Changing the Culture of Tobacco Dependence Treatment Among Not Only Patients, But Also Prescribers. Mayo Clin Proc. 2021 Sep;96(9):2495. doi: 10.1016/j.mayocp.2021.07.010. No abstract available. PMID 34481605
- [Derived] Ebbert J, Jimenez-Ruiz C, Dutro MP, Fisher M, Li J, Hays JT. Frequently Reported Adverse Events With Smoking Cessation Medications: Post Hoc Analysis of a Randomized Trial. Mayo Clin Proc. 2021 Jul;96(7):1801-1811. doi: 10.1016/j.mayocp.2020.10.046. Epub 2021 Jun 8. PMID 34112520
- [Derived] Beard E, Jackson SE, Anthenelli RM, Benowitz NL, Aubin LS, McRae T, Lawrence D, Russ C, Krishen A, Evins AE, West R. Estimation of risk of neuropsychiatric adverse events from varenicline, bupropion and nicotine patch versus placebo: secondary analysis of results from the EAGLES trial using Bayes factors. Addiction. 2021 Oct;116(10):2816-2824. doi: 10.1111/add.15440. Epub 2021 Apr 22. PMID 33885203
- [Derived] Correa JB, Lawrence D, McKenna BS, Gaznick N, Saccone PA, Dubrava S, Doran N, Anthenelli RM. Psychiatric Comorbidity and Multimorbidity in the EAGLES Trial: Descriptive Correlates and Associations With Neuropsychiatric Adverse Events, Treatment Adherence, and Smoking Cessation. Nicotine Tob Res. 2021 Aug 29;23(10):1646-1655. doi: 10.1093/ntr/ntab056. PMID 33788933
- [Derived] Nollen NL, Ahluwalia JS, Sanderson Cox L, Okuyemi K, Lawrence D, Samuels L, Benowitz NL. Assessment of Racial Differences in Pharmacotherapy Efficacy for Smoking Cessation: Secondary Analysis of the EAGLES Randomized Clinical Trial. JAMA Netw Open. 2021 Jan 4;4(1):e2032053. doi: 10.1001/jamanetworkopen.2020.32053. PMID 33464316
- [Derived] Evins AE, West R, Benowitz NL, Russ C, Lawrence D, McRae T, Maravic MC, Heffner JL, Anthenelli RM. Efficacy and Safety of Pharmacotherapeutic Smoking Cessation Aids in Schizophrenia Spectrum Disorders: Subgroup Analysis of EAGLES. Psychiatr Serv. 2021 Jan 1;72(1):7-15. doi: 10.1176/appi.ps.202000032. Epub 2020 Nov 3. PMID 33138708
- [Derived] Ayers CR, Heffner JL, Russ C, Lawrence D, McRae T, Evins AE, Anthenelli RM. Efficacy and safety of pharmacotherapies for smoking cessation in anxiety disorders: Subgroup analysis of the randomized, active- and placebo-controlled EAGLES trial. Depress Anxiety. 2020 Mar;37(3):247-260. doi: 10.1002/da.22982. Epub 2019 Dec 18. PMID 31850603
- [Derived] Heffner JL, Evins AE, Russ C, Lawrence D, Ayers CR, McRae T, Aubin LS, Krishen A, West R, Anthenelli RM. Safety and efficacy of first-line smoking cessation pharmacotherapies in bipolar disorders: Subgroup analysis of a randomized clinical trial. J Affect Disord. 2019 Sep 1;256:267-277. doi: 10.1016/j.jad.2019.06.008. Epub 2019 Jun 3. PMID 31195244
- [Derived] Anthenelli RM, Gaffney M, Benowitz NL, West R, McRae T, Russ C, Lawrence D, St Aubin L, Krishen A, Evins AE. Predictors of Neuropsychiatric Adverse Events with Smoking Cessation Medications in the Randomized Controlled EAGLES Trial. J Gen Intern Med. 2019 Jun;34(6):862-870. doi: 10.1007/s11606-019-04858-2. Epub 2019 Mar 7. PMID 30847828
- [Derived] West R, Evins AE, Benowitz NL, Russ C, McRae T, Lawrence D, St Aubin L, Krishen A, Maravic MC, Anthenelli RM. Factors associated with the efficacy of smoking cessation treatments and predictors of smoking abstinence in EAGLES. Addiction. 2018 Aug;113(8):1507-1516. doi: 10.1111/add.14208. Epub 2018 Mar 30. PMID 29508470
- [Derived] Anthenelli RM, Benowitz NL, West R, St Aubin L, McRae T, Lawrence D, Ascher J, Russ C, Krishen A, Evins AE. Neuropsychiatric safety and efficacy of varenicline, bupropion, and nicotine patch in smokers with and without psychiatric disorders (EAGLES): a double-blind, randomised, placebo-controlled clinical trial. Lancet. 2016 Jun 18;387(10037):2507-20. doi: 10.1016/S0140-6736(16)30272-0. Epub 2016 Apr 22. PMID 27116918

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 11,186 participants were screened for participation in the study, of which 3042 participants were considered to be screen failures, leaving 8144 participants eligible for study participation (efficacy population). 86 participants (1.1%) did not receive study drug. A total of 8058 participants received study drug (safety population).
Pre-assignment Details: Participants were classified into 2 cohorts: participants without diagnosis of psychiatric disorder and participants with a stable diagnosis of psychiatric disorder confirmed by the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders (SCID) 4th edition conducted at screening.
Groups:
- Varenicline: Participants were randomized to 1 of the 3 active dosing groups that took active medication of either varenicline, bupropion, NRT in this triple-dummy design. Participants in this arm received varenicline titrated to the full dose during the first week in the following manner: 0.5 mg daily once (QD) x 3 days, 0.5 mg twice daily (BID) x 4 days, then 1 mg BID for 11 weeks. They also received placebo bupropion and NRT patch, dosed in the same manner as the active medication.
- Bupropion: Participants were randomized to 1 of the 3 active dosing groups that took active medication of either varenicline, bupropion, NRT in this triple-dummy design. Participants in this arm received bupropion 150 mg QD x 3 days and taken 150 mg BID for the remainder of the treatment period (11 weeks and 4 days). They also received placebo varenicline and NRT patch, dosed in the same manner as the active medication.
- NRT Patch: Participants were randomized to 1 of the 3 active dosing groups that took active medication of either varenicline, bupropion, NRT in this triple-dummy design. Participants in this arm received NRT started active dosing the morning of the Week 1 visit and received a 21 mg transdermal patch per day x 7 weeks, followed by a 14 mg transdermal patch per day x 2 weeks, and then a 7 mg transdermal patch x 2 weeks for a total of 11 weeks of treatment. They also received placebo varenicline and bupropion, dosed in the same manner as active medication.
- Placebo: Participants received matching placebo for varenicline, bupropion, and NRT in this triple-dummy design, and followed the same titration and dosing schedule as for the active treatments noted above.
Period: Overall Study
Arm/Group | Varenicline | Bupropion | NRT Patch | Placebo
Started | 2037 | 2034 | 2038 | 2035
Randomized and Treated | 2016 | 2006 | 2022 | 2014
Completed | 1598 | 1586 | 1557 | 1552
Not Completed | 439 | 448 | 481 | 483
Not completed — Other reason | 41 | 30 | 36 | 33
Not completed — No longer meets eligibility criteria | 4 | 8 | 6 | 5
Not completed — Protocol Violation | 4 | 2 | 5 | 5
Not completed — Pregnancy | 1 | 0 | 0 | 1
Not completed — Insufficient clinical response | 4 | 4 | 14 | 13
Not completed — No longer willing to participate | 195 | 218 | 224 | 248
Not completed — Lost to Follow-up | 135 | 126 | 144 | 127
Not completed — Medication error | 0 | 1 | 0 | 1
Not completed — Adverse event (study drug) | 25 | 21 | 26 | 17
Not completed — Adverse event (study drug unrelated) | 9 | 7 | 9 | 9
Not completed — Death | 0 | 3 | 1 | 3
Not completed — Randomized but not treated | 21 | 28 | 16 | 21

BASELINE CHARACTERISTICS:
Population: The safety analysis population contained all treated participants i.e. who received at least one partial dose of study medication.
Groups:
- Varenicline 1.0 mg BID: Participants were randomized to 1 of the 3 active dosing groups that took active medication of either varenicline, bupropion, NRT in this triple-dummy design. Participants in this arm received varenicline titrated to the full dose during the first week in the following manner: 0.5 mg QD x 3 days, 0.5 mg BID x 4 days, then 1 mg BID for 11 weeks. They also received placebo bupropion and NRT patch, dosed in the same manner as the active medication.
- Total: Total of all reporting groups
Arm/Group | Varenicline 1.0 mg BID | Bupropion | NRT Patch | Placebo | Total
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014 | 8058
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.5 (12.4) | 46.3 (12.6) | 46.8 (12.2) | 46.4 (12.2) | 46.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1114 | 1116 | 1141 | 1138 | 4509
  Male | 902 | 890 | 881 | 876 | 3549

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Neuropsychiatric (NPS) Adverse Events (AE) - the Primary Study Endpoint
Description: The primary safety endpoint is the occurrence of at least one treatment emergent "severe" adverse event of anxiety, depression, feeling abnormal, or hostility and/or the occurrence of at least one treatment emergent "moderate" or "severe" adverse event of: agitation, aggression, delusions, hallucinations, homicidal ideation, mania, panic, paranoia, psychosis, suicidal ideation, suicidal behavior, or completed suicide.
Time Frame: Treatment emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: The safety dataset included all participants who had received at least one partial dose of study medication (N=8058) and was used to analyze all safety endpoints.
Measure: Number; unit: percentage of participants
Groups:
- Bupropion 150 mg BID: Participants were randomized to 1 of the 3 active dosing groups that took active medication of either varenicline, bupropion, NRT in this triple-dummy design. Participants in this arm received bupropion 150 mg QD x 3 days and taken 150 mg BID for the remainder of the treatment period (11 weeks and 4 days). They also received placebo varenicline and NRT patch, dosed in the same manner as the active medication.
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
percentage of participants
  Non-psychiatric cohort (N= 990, 989, 1006, 999) | 1.3 | 2.2 | 2.5 | 2.4
  Psychiatric cohort (N= 1026, 1017, 1016, 1015) | 6.5 | 6.7 | 5.2 | 4.9
  Overall (N= 2016, 2006, 2022, 2014) | 4.0 | 4.5 | 3.9 | 3.7
Statistical Analysis 1: Comparison: Varenicline 1.0 mg BID vs Bupropion 150 mg BID vs NRT Patch vs Placebo; The reduced (final) statistical model included treatment group, cohort and region, plus the 2-way interaction of treatment by cohort. Other interactions not included due to lack of significance. Region reduced to 2-level to address event sparseness issue; Test type: Superiority or Other; p = 0.0652, Regression, Linear — An interaction between treatment and cohort was considered significant at 10% level. No multiplicity adjustments were utilized; A generalized linear regression analysis based on the safety analysis set was used to evaluate incidence of NPS AE as the primary analysis

2. Primary Outcome: Estimated NPS AE Rate (%), by Cohort
Description: The primary safety endpoint is the occurrence of at least one treatment emergent "severe" adverse event of anxiety, depression, feeling abnormal, or hostility and/or the occurrence of at least one treatment emergent "moderate" or "severe" adverse event of: agitation, aggression, delusions, hallucinations, homicidal ideation, mania, panic, paranoia, psychosis, suicidal ideation, suicidal behavior, or completed suicide. Estimated NPS AE rate (%) was calculated based on least-squares means analysis.
Time Frame: Treatment emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
percentage of participants
  Non-psychiatric cohort (N=3984) | 1.25 [0.60 to 1.90] | 2.44 [1.52 to 3.36] | 2.31 [1.37 to 3.25] | 2.52 [1.58 to 3.46]
  Psychiatric cohort (N= 4074) | 6.42 [4.91 to 7.93] | 6.62 [5.09 to 8.15] | 5.20 [3.84 to 6.56] | 4.83 [3.51 to 6.16]
Statistical Analysis 1: Comparison: Varenicline 1.0 mg BID vs Placebo; Non-psychiatric cohort; Test type: Superiority or Other; Regression, Linear; Risk Difference (RD) = -1.28, 95% CI 2-sided [-2.40 to -0.15] — Risk difference for varenicline versus placebo from estimation model
Statistical Analysis 2: Comparison: Bupropion 150 mg BID vs Placebo; Non-psychiatric cohort; Test type: Superiority or Other; Regression, Linear; Risk Difference (RD) = -0.08, 95% CI 2-sided [-1.37 to 1.21] — Risk difference for bupropion 150 mg BID versus placebo from estimation model
Statistical Analysis 3: Comparison: NRT Patch vs Placebo; Non-psychiatric cohort; Test type: Superiority or Other; Regression, Linear; Risk Difference (RD) = -0.21, 95% CI 2-sided [-1.54 to 1.12] — Risk difference for NRT versus placebo from estimation model
Statistical Analysis 4: Comparison: Varenicline 1.0 mg BID vs Placebo; Psychiatric cohort; Test type: Superiority or Other; Regression, Linear; Risk Difference (RD) = 1.59, 95% CI 2-sided [-0.42 to 3.59] — Risk difference for varenicline versus placebo from estimation model
Statistical Analysis 5: Comparison: Bupropion 150 mg BID vs Placebo; Psychiatric cohort; Test type: Superiority or Other; Regression, Linear; Risk Difference (RD) = 1.78, 95% CI 2-sided [-0.24 to 3.81] — Risk difference for bupropion 150 mg BID versus placebo from estimation model
Statistical Analysis 6: Comparison: NRT Patch vs Placebo; Psychiatric cohort; Test type: Superiority or Other; Regression, Linear; Risk Difference (RD) = 0.37, 95% CI 2-sided [-1.53 to 2.26] — Risk difference for NRT versus placebo from estimation model

3. Secondary Outcome: Occurrence of the Components of the NPS AE Primary Endpoint, Non-psychiatric History Cohort
Description: The safety endpoint is the occurrence of at least one treatment emergent "severe" adverse event of anxiety, depression, feeling abnormal, or hostility and/or the occurrence of at least one treatment emergent "moderate" or "severe" adverse event of: agitation, aggression, delusions, hallucinations, homicidal ideation, mania, panic, paranoia, psychosis, suicidal ideation, suicidal behavior, or completed suicide. Each of these 16 components is reported below.
Time Frame: Treatment emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 990 | 989 | 1006 | 999
participants
  Anxiety (severe) | 0 | 1 | 0 | 3
  Depression (severe) | 1 | 0 | 0 | 0
  Feeling abnormal (severe only) | 0 | 0 | 0 | 0
  Hostility (severe) | 0 | 1 | 1 | 0
  Agitation (moderate and severe) | 10 | 11 | 19 | 11
  Aggression (moderate and severe) | 3 | 3 | 2 | 3
  Delusions (moderate and severe) | 0 | 0 | 1 | 0
  Hallucinations (moderate and severe) | 1 | 0 | 0 | 0
  Mania (moderate and severe) | 0 | 1 | 2 | 2
  Panic (moderate and severe) | 0 | 4 | 1 | 3
  Paranoia (moderate and severe) | 0 | 1 | 0 | 0
  Psychosis (moderate and severe) | 0 | 0 | 1 | 0
  Homicidal ideation (moderate and severe) | 0 | 0 | 1 | 0
  Suicidal behavior (moderate and severe) | 0 | 1 | 1 | 0
  Suicidal ideation (moderate and severe) | 0 | 1 | 2 | 3
  Suicide (moderate and severe) | 0 | 0 | 0 | 1

4. Secondary Outcome: Occurrence of the Components of the NPS AE Primary Endpoint, Psychiatric History Cohort
Description: as for outcome 3
Time Frame: Treatment emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 1026 | 1017 | 1016 | 1015
participants
  Anxiety (severe) | 5 | 4 | 6 | 2
  Depression (severe) | 6 | 4 | 7 | 6
  Feeling abnormal (severe only) | 0 | 1 | 0 | 0
  Hostility (severe) | 0 | 0 | 0 | 0
  Agitation (moderate and severe) | 25 | 29 | 21 | 22
  Aggression (moderate and severe) | 14 | 9 | 7 | 8
  Delusions (moderate and severe) | 1 | 1 | 1 | 0
  Hallucinations (moderate and severe) | 5 | 4 | 2 | 2
  Mania (moderate and severe) | 7 | 9 | 3 | 6
  Panic (moderate and severe) | 7 | 16 | 13 | 7
  Paranoia (moderate and severe) | 1 | 0 | 0 | 2
  Psychosis (moderate and severe) | 4 | 2 | 3 | 1
  Homicidal ideation (moderate and severe) | 0 | 0 | 0 | 0
  Suicidal behavior (moderate and severe) | 1 | 1 | 0 | 1
  Suicidal ideation (moderate and severe) | 5 | 2 | 3 | 2
  Suicide (moderate and severe) | 0 | 0 | 0 | 0

5. Secondary Outcome: Occurrence of the Components of NPS AE Primary Endpoint (Overall)
Description: The NPS AE composite results (as previously described) are for the two cohorts combined and are presented below.
Time Frame: Treatment emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
participants
  Anxiety | 5 | 5 | 6 | 5
  Depression | 7 | 4 | 7 | 6
  Feeling Abnormal | 0 | 1 | 0 | 0
  Hostility | 0 | 1 | 1 | 0
  Agitation | 35 | 40 | 40 | 33
  Aggression | 17 | 12 | 9 | 11
  Delusions | 1 | 1 | 2 | 0
  Hallucination | 6 | 4 | 2 | 2
  Mania | 7 | 10 | 5 | 8
  Panic Disorder | 7 | 20 | 14 | 10
  Paranoia | 1 | 1 | 0 | 2
  Psychosis | 4 | 2 | 4 | 1
  Homicidal Ideation | 0 | 0 | 1 | 0
  Suicidal Behavior | 1 | 2 | 1 | 1
  Suicidal Ideation | 5 | 3 | 5 | 5
  Suicide | 0 | 0 | 0 | 1

6. Secondary Outcome: Occurrence of Severe-only NPS AEs in the Primary Endpoint, by Cohort
Description: The primary safety endpoint is the occurrence of at least one treatment emergent "severe" adverse event of anxiety, depression, feeling abnormal, or hostility and/or the occurrence of at least one treatment emergent "moderate" or "severe" adverse event of: agitation, aggression, delusions, hallucinations, homicidal ideation, mania, panic, paranoia, psychosis, suicidal ideation, suicidal behavior, or completed suicide. Only those events rated as severe are reported; this excludes any moderate events in the primary NPS AE endpoint.
Time Frame: Treatment emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
percentage of participants
  Non-psychiatric cohort (N= 990, 989, 1006, 999) | 0.1 | 0.4 | 0.3 | 0.5
  Psychiatric cohort (N= 1026, 1017, 1016, 1015) | 1.4 | 1.4 | 1.4 | 1.3
  Overall (N= 2016, 2006, 2022, 2014) | 0.7 | 0.9 | 0.8 | 0.9

7. Secondary Outcome: Occurrence of the Components of the Observed Severe-only NPS AE Primary Endpoint, Non-psychiatric History Cohort
Description: The safety endpoint is the occurrence of at least one treatment emergent "severe" adverse event of anxiety, depression, feeling abnormal, or hostility and/or the occurrence of at least one treatment emergent "moderate" or "severe" adverse event of: agitation, aggression, delusions, hallucinations, homicidal ideation, mania, panic, paranoia, psychosis, suicidal ideation, suicidal behavior, or completed suicide. Only those events rated as severe are reported; this excludes any moderate events in the primary NPS AE endpoint.
Time Frame: Treatment emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 990 | 989 | 1006 | 999
participants
  Anxiety | 0 | 1 | 0 | 3
  Depression | 1 | 0 | 0 | 0
  Feeling abnormal | 0 | 0 | 0 | 0
  Hostility | 0 | 1 | 1 | 0
  Agitation | 0 | 0 | 2 | 0
  Aggression | 1 | 1 | 0 | 0
  Delusions | 0 | 0 | 0 | 0
  Hallucinations | 0 | 0 | 0 | 0
  Mania | 0 | 0 | 0 | 0
  Panic | 0 | 1 | 1 | 1
  Paranoia | 0 | 0 | 0 | 0
  Psychosis | 0 | 0 | 0 | 0
  Homicidal ideation | 0 | 0 | 0 | 0
  Suicidal behavior | 0 | 1 | 0 | 0
  Suicidal ideation | 0 | 0 | 0 | 1
  Suicide | 0 | 0 | 0 | 1

8. Secondary Outcome: Occurrence of the Components of the Observed Severe-only NPS AE Primary Endpoint, Psychiatric History Cohort
Description: as for outcome 7
Time Frame: Treatment emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 1026 | 1017 | 1016 | 1015
participants
  Anxiety | 5 | 4 | 6 | 2
  Depression | 6 | 4 | 7 | 6
  Feeling abnormal | 0 | 1 | 0 | 0
  Hostility | 0 | 0 | 0 | 0
  Agitation | 1 | 1 | 4 | 2
  Aggression | 1 | 1 | 0 | 1
  Delusions | 0 | 0 | 0 | 0
  Hallucinations | 0 | 1 | 0 | 0
  Mania | 2 | 1 | 0 | 0
  Panic | 0 | 1 | 0 | 1
  Paranoia | 0 | 0 | 0 | 0
  Psychosis | 0 | 1 | 1 | 0
  Homicidal ideation | 0 | 0 | 0 | 0
  Suicidal behavior | 1 | 1 | 0 | 1
  Suicidal ideation | 1 | 0 | 1 | 0
  Suicide | 0 | 0 | 0 | 0

9. Secondary Outcome: Occurrence of the Components of Severe-only NPS AE Endpoint (Overall)
Description: The NPS AE endpoint was the occurrence of at least 1 treatment-emergent "severe" AE of anxiety, depression, feeling abnormal, or hostility and/or the occurrence of at least 1 treatment-emergent "severe" AE of agitation, aggression, delusions, hallucinations, homicidal ideation, mania, panic, paranoia, psychosis, suicidal ideation, suicidal behavior, or completed suicide. Only those events rated as severe are reported; this excludes any moderate events in the primary NPS AE endpoint.
Time Frame: Treatment emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
participants
  Anxiety | 5 | 5 | 6 | 5
  Depression | 7 | 4 | 7 | 6
  Feeling Abnormal | 0 | 1 | 0 | 0
  Hostility | 0 | 1 | 1 | 0
  Agitation | 1 | 1 | 6 | 2
  Aggression | 2 | 2 | 0 | 1
  Delusions | 0 | 0 | 0 | 0
  Hallucination | 0 | 1 | 0 | 0
  Mania | 2 | 1 | 0 | 0
  Panic Disorder | 0 | 2 | 1 | 2
  Paranoia | 1 | 1 | 0 | 2
  Psychosis | 4 | 2 | 4 | 1
  Suicidal Behavior | 1 | 2 | 0 | 1
  Suicidal Ideation | 1 | 0 | 1 | 0
  Suicide | 0 | 0 | 0 | 1
  Homicidal Ideation | 0 | 0 | 1 | 0

10. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Total Score, Non-psychiatric History Cohort
Description: The HADS is a subject self-reporting scale completed in person at clinic visits at Baseline and Weeks 1 through 6, 8, 10, 12, 13, 16, 20, and 24. It contains 14 individual item responses ranging in increasing severity from 0 (normal) to 3 (most severe) for a total range of 0 to 42. Of the 14 items, 7 assess anxiety and 7 assess depression, providing 2 subscales with ranges of 0 to 21. For each subscale, 0 to 7 is considered normal, while 15 to 21 represents severe symptoms.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 990 | 989 | 1006 | 999
Units on a scale
  Week 1 (N= 984, 972, 989, 992) | 3.26 (3.92) | 3.58 (4.25) | 3.06 (3.87) | 3.38 (4.20)
  Week 2 (N= 961, 954, 963, 970) | 2.91 (3.86) | 3.07 (3.96) | 2.84 (3.85) | 3.20 (4.25)
  Week 3 (N= 935, 930, 936, 941) | 2.61 (3.85) | 2.64 (3.82) | 2.63 (3.93) | 2.77 (3.94)
  Week 4 (N= 923, 916, 934, 923) | 2.40 (3.66) | 2.36 (3.57) | 2.46 (3.80) | 2.77 (4.21)
  Week 5 (N= 911, 897, 906, 902) | 2.29 (3.51) | 2.24 (3.52) | 2.32 (3.86) | 2.48 (3.92)
  Week 6 (N= 899, 893, 909, 897) | 2.23 (3.56) | 2.18 (3.57) | 2.40 (3.87) | 2.48 (3.97)
  Week 8 (N= 868, 861, 877, 877) | 2.17 (3.60) | 2.16 (3.70) | 2.28 (3.60) | 2.64 (4.29)
  Week 10 (N= 853, 844, 852, 846) | 2.29 (3.89) | 1.96 (3.24) | 2.33 (3.80) | 2.57 (4.41)
  Week 12 (N= 772, 768, 750, 742) | 2.07 (3.48) | 1.83 (3.21) | 2.01 (3.51) | 2.46 (4.10)
  Week 13 (N= 797, 796, 789, 807) | 2.11 (3.74) | 1.85 (3.22) | 2.01 (3.47) | 2.38 (4.27)
  Week 16 (N= 784, 797, 775, 789) | 2.05 (3.47) | 1.90 (3.43) | 2.09 (3.61) | 2.34 (3.98)
  Week 20 (N= 771, 785, 762, 772) | 2.10 (3.54) | 1.93 (3.36) | 1.97 (3.53) | 2.31 (4.15)
  Week 24 (N= 758, 748, 737, 758) | 2.01 (3.49) | 1.87 (3.47) | 2.01 (3.45) | 2.25 (4.04)

11. Secondary Outcome: HADS Total Score, Psychiatric History Cohort
Description: as for outcome 10
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 1026 | 1017 | 1016 | 1015
Units on a scale
  Week 1 (N= 1026, 1017, 1015, 1015) | 6.76 (6.14) | 7.58 (6.87) | 6.82 (6.33) | 6.70 (5.94)
  Week 2 (N= 1005, 1004, 996, 995) | 6.42 (6.36) | 6.99 (6.47) | 6.64 (6.55) | 6.42 (6.17)
  Week 3 (N= 947, 961, 945, 926) | 5.99 (6.21) | 6.51 (6.39) | 6.30 (6.55) | 6.02 (6.10)
  Week 4 (N= 935, 938, 929, 908) | 5.87 (6.39) | 6.36 (6.55) | 6.16 (6.51) | 6.04 (6.31)
  Week 5 (N= 918, 918, 914, 895) | 5.58 (6.32) | 6.03 (6.41) | 5.82 (6.44) | 5.80 (6.31)
  Week 6 (N= 917, 914, 912, 874) | 5.39 (6.14) | 5.87 (6.41) | 5.62 (6.22) | 5.75 (6.26)
  Week 8 (N= 887, 893, 878, 859) | 5.43 (6.24) | 5.96 (6.68) | 5.63 (6.36) | 5.63 (6.26)
  Week 10 (N= 864, 865, 864, 823) | 5.38 (6.35) | 5.72 (6.50) | 5.64 (6.30) | 5.55 (6.38)
  Week 12 (N= 790, 803, 798, 749) | 5.17 (6.09) | 5.66 (6.63) | 5.44 (6.30) | 5.42 (6.13)
  Week 13 (N= 813, 812, 814, 763) | 5.06 (6.11) | 5.44 (6.54) | 5.36 (6.20) | 5.09 (5.96)
  Week 16 (N= 795, 805, 791, 748) | 5.26 (6.35) | 5.62 (6.68) | 5.44 (6.34) | 5.37 (6.38)
  Week 20 (N= 784, 784, 763, 737) | 5.17 (6.02) | 5.54 (6.44) | 5.46 (6.18) | 5.26 (6.22)
  Week 24 (N= 770, 764, 758, 729) | 5.21 (6.27) | 5.69 (6.64) | 5.57 (6.32) | 5.04 (5.97)

12. Secondary Outcome: HADS Total Score (Overall)
Description: as for outcome 10
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2021 | 2014
Units on a scale
  Week 1 (N= 1989, 1976, 1985, 1987) | 5.03 (5.45) | 5.61 (6.07) | 4.95 (5.58) | 5.05 (5.41)
  Week 2 (N= 1938, 1937, 1931, 1929) | 4.68 (5.55) | 5.06 (5.73) | 4.74 (5.70) | 4.80 (5.53)
  Week 3 (N= 1882, 1891, 1881, 1867) | 4.31 (5.44) | 4.60 (5.63) | 4.48 (5.71) | 4.38 (5.37)
  Week 4 (N= 1858, 1854, 1863, 1831) | 4.15 (5.50) | 4.39 (5.65) | 4.31 (5.64) | 4.39 (5.60)
  Week 5 (N= 1829, 1815, 1820, 1797) | 3.94 (5.37) | 4.16 (5.52) | 4.08 (5.59) | 4.14 (5.51)
  Week 6 (N= 1816, 1807, 1821, 1771) | 3.82 (5.27) | 4.05 (5.52) | 4.01 (5.42) | 4.09 (5.48)
  Week 8 (N= 1755, 1754, 1755, 1736) | 3.82 (5.36) | 4.10 (5.75) | 3.96 (5.43) | 4.12 (5.56)
  Week 10 (N= 1717, 1709, 1716, 1669) | 3.85 (5.49) | 3.86 (5.48) | 4.00 (5.47) | 4.04 (5.67)
  Week 12 (N= 1562, 1571, 1548, 1491) | 3.64 (5.21) | 3.79 (5.58) | 3.78 (5.42) | 3.95 (5.42)
  Week 13 (N= 1610, 1608, 1603, 1570) | 3.60 (5.29) | 3.66 (5.47) | 3.71 (5.32) | 3.70 (5.34)
  Week 16 (N= 1579, 1602, 1566, 1537) | 3.67 (5.37) | 3.77 (5.63) | 3.78 (5.44) | 3.82 (5.50)
  Week 20 (N= 1555, 1569, 1525, 1509) | 3.65 (5.18) | 3.73 (5.44) | 3.72 (5.33) | 3.75 (5.47)
  Week 24 (N= 1528, 1512, 1495, 1487) | 3.62 (5.33) | 3.80 (5.64) | 3.82 (5.41) | 3.62 (5.27)

13. Secondary Outcome: Positive Responses for Suicidal Behavior and/or Ideation by Columbia Suicide Severity Rating Scale (C-SSRS) - Non-psychiatric History Cohort
Description: The C-SSRS is a semi-structured interview designed to evaluate an individual's degree of suicidal ideation, preparatory acts or behavior to actual attempt, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent". Answers at screening are for lifetime history. Answers for all other visits are since last visit.The scale is also used to record any completed suicides.
Time Frame: Lifetime, Baseline and Treatment-Emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Number; unit: participants with positive responses
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 990 | 989 | 1006 | 999
participants with positive responses
  Suicidal Behavior (Screening lifetime) | 6 | 9 | 7 | 6
  Suicidal Ideation (Screening lifetime) | 48 | 43 | 50 | 49
  Suicidal Behavior (Baseline) | 0 | 0 | 0 | 0
  Suicidal Ideation (Baseline) | 0 | 1 | 0 | 1
  Suicidal Behavior (treatment emergent 12 weeks) | 0 | 0 | 1 | 1
  Suicidal Ideation (treatment emergent 12 weeks) | 7 | 4 | 3 | 6

14. Secondary Outcome: Positive Responses for Suicidal Behavior and/or Ideation by Columbia Suicide Severity Rating Scale (C-SSRS) - Psychiatric History Cohort
Description: The C-SSRS is a semi-structured interview designed to evaluate an individual's degree of suicidal ideation, preparatory acts or behavior to actual attempt, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent". Answers at screening are for lifetime history. Answers for all other visits are since last visit. The scale is also used to record any completed suicides.
Time Frame: Lifetime, Baseline and Treatment-Emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Number; unit: participants with positive responses
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 1026 | 1017 | 1016 | 1015
participants with positive responses
  Suicidal Behavior (Screening lifetime) | 137 | 143 | 111 | 123
  Suicidal Ideation (Screening lifetime) | 338 | 357 | 333 | 349
  Suicidal Behavior (Baseline) | 0 | 0 | 0 | 1
  Suicidal Ideation (Baseline) | 6 | 5 | 2 | 3
  Suicidal Behavior (treatment emergent 12 weeks) | 0 | 1 | 0 | 2
  Suicidal Ideation (treatment emergent 12 weeks) | 27 | 15 | 20 | 25

15. Secondary Outcome: Positive Responses for Suicidal Behavior and/or Ideation by Columbia Suicide Severity Rating Scale (C-SSRS) - Overall
Description: as for outcome 14
Time Frame: Lifetime, Baseline and Treatment-Emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Population: as for outcome 1
Measure: Number; unit: participants with positive responses
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
participants with positive responses
  Suicidal Behavior (Screening lifetime) | 143 | 152 | 118 | 129
  Suicidal Ideation (Screening lifetime) | 386 | 400 | 383 | 398
  Suicidal Behavior (Baseline) | 0 | 0 | 0 | 1
  Suicidal Ideation (Baseline) | 6 | 6 | 2 | 4
  Suicidal Behavior (treatment emergent 12 weeks) | 0 | 1 | 1 | 3
  Suicidal Ideation (treatment emergent 12 weeks) | 34 | 19 | 23 | 31

16. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I), "No Change" Rating by Visit
Description: The CGI-I is a clinician rated instrument that measures change in participant's psychiatric condition (or lack thereof in the stratum without psychiatric disorders) on a 7 point scale ranging from 1 (very much improved) to 7 (very much worse), with 4 = no change. The ratings were applicable even to those without psychiatric diagnoses (eg, those with no psychiatric symptoms would be rated as "normal, not at all ill" on the CGI-S at baseline and assuming no psychiatric symptoms emerge during the trial, would be rated as "no change" on the CGI-I at follow-up visits). For those participants with a psychiatric diagnosis, the clinician should rate the severity of the mental illness with respect to the clinician's experience with the psychiatric population to which the participant belongs.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 2016 | 2006 | 2022 | 2014
percentage of participants
  Week 1 (N= 1986, 1974, 1986, 1982) | 94.2 | 93.2 | 94.6 | 95.1
  Week 2 (N= 1934, 1936, 1927, 1926) | 90.8 | 90.8 | 90.5 | 91.2
  Week 3 (N= 1880, 1892, 1880, 1863) | 88.3 | 89.8 | 88.7 | 87.9
  Week 4 (N= 1860, 1856, 1858, 1834) | 86.6 | 88.0 | 87.1 | 86.3
  Week 5 (N= 1828, 1816, 1822, 1802) | 85.7 | 86.5 | 85.5 | 85.4
  Week 6 (N= 1816, 1808, 1820, 1773) | 85.2 | 86.5 | 85.1 | 84.1
  Week 8 (N= 1758, 1756, 1755, 1738) | 82.4 | 83.6 | 82.8 | 81.9
  Week 10 (N= 1717, 1707, 1715, 1675) | 80.6 | 81.7 | 80.4 | 79.2
  Week 12 (N= 1558, 1572, 1540, 1492) | 72.9 | 75.1 | 72.2 | 71.3
  Week 13 (N= 1612, 16081602, 1575) | 75.9 | 76.7 | 75.2 | 74.9
  Week 16 (N= 1586, 1606, 1568, 1541) | 74.2 | 76.7 | 73.9 | 73.4
  Week 20 (N= 1563, 1573, 1523, 1510) | 73.4 | 75.0 | 72.2 | 71.7
  Week 24 (N= 1533, 1515, 1499, 1497) | 71.8 | 72.3 | 71.1 | 71.1

17. Secondary Outcome: CO-Confirmed Continuous Abstinence for Weeks 9 Through 12, Non-psychiatric History Cohort
Description: A responder to this endpoint requires the answer "no" to both questions 1 and 2 on the Nicotine Use Inventory at every visit from Week 9 to Week 12 (inclusive).
Time Frame: Week 9 through Week 12
Population: The full analysis set was defined under the intent-to-treat (ITT) principle as all randomized participants (N=8144) and was used for all efficacy endpoints.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 1005 | 1001 | 1013 | 1009
percentage of participants | 38.0 | 26.1 | 26.4 | 13.7
Statistical Analysis 1: Comparison: Varenicline 1.0 mg BID vs Placebo; The analysis was done using a logistic regression with terms treatment, cohort, region, treatment by cohort interaction, and region by cohort interaction. Region reduced to 2-level for consistency with primary safety model; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 4.00, 95% CI 2-sided [3.20 to 5.00]
Statistical Analysis 2: Comparison: Bupropion 150 mg BID vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.80 to 2.85]
Statistical Analysis 3: Comparison: NRT Patch vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.30, 95% CI 2-sided [1.83 to 2.90]

18. Secondary Outcome: CO-Confirmed Continuous Abstinence for Weeks 9 Through 12, Psychiatric History Cohort
Description: as for outcome 17
Time Frame: Week 9 through Week 12
Population: The full analysis set was defined under the ITT principle as all randomized participants (N=8144) and was used for all efficacy endpoints.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 1032 | 1033 | 1025 | 1026
percentage of participants | 29.2 | 19.3 | 20.4 | 11.4
Statistical Analysis 1: Comparison: Varenicline 1.0 mg BID vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 3.24, 95% CI 2-sided [2.56 to 4.11]
Statistical Analysis 2: Comparison: Bupropion 150 mg BID vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.46 to 2.39]
Statistical Analysis 3: Comparison: NRT Patch vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.56 to 2.55]

19. Secondary Outcome: CO-Confirmed Continuous Abstinence for Weeks 9 Through 12 (Overall)
Description: as for outcome 17
Time Frame: Week 9 through Week 12
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 2037 | 2034 | 2038 | 2035
percentage of participants | 33.5 | 22.6 | 23.4 | 12.5
Statistical Analysis 1: Comparison: Varenicline 1.0 mg BID vs Placebo; The analysis was done using a logistic regression with terms treatment and region. Region reduced to 2-level for consistency with primary safety model; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 3.61, 95% CI 2-sided [3.07 to 4.24]
Statistical Analysis 2: Comparison: Bupropion 150 mg BID vs Placebo; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.07, 95% CI 2-sided [1.75 to 2.45]
Statistical Analysis 3: Comparison: NRT Patch vs Placebo; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.82 to 2.54]

20. Secondary Outcome: CO-confirmed Continuous Abstinence From Week 9 Through Week 24, Non-psychiatric History Cohort
Description: A responder to this endpoint requires the answer "no" to both questions 1 and 2 on the Nicotine Use Inventory at every visit from Week 9 to Week 24 (inclusive).
Time Frame: Week 9 through Week 24
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 1005 | 1001 | 1013 | 1009
percentage of participants | 25.5 | 18.8 | 18.5 | 10.5
Statistical Analysis 1: Comparison: Varenicline 1.0 mg BID vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.99, 95% CI 2-sided [2.33 to 3.83]
Statistical Analysis 2: Comparison: Bupropion 150 mg BID vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.54 to 2.59]
Statistical Analysis 3: Comparison: NRT Patch vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 1.96, 95% CI 2-sided [1.51 to 2.54]

21. Secondary Outcome: CO-confirmed Continuous Abstinence From Week 9 Through Week 24, Psychiatric History Cohort
Description: as for outcome 20
Time Frame: Week 9 through Week 24
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 1032 | 1033 | 1025 | 1026
percentage of participants | 18.3 | 13.7 | 13.0 | 8.3
Statistical Analysis 1: Comparison: Varenicline 1.0 mg BID vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.50, 95% CI 2-sided [1.90 to 3.29]
Statistical Analysis 2: Comparison: Bupropion 150 mg BID vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.33 to 2.36]
Statistical Analysis 3: Comparison: NRT Patch vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.24 to 2.20]

22. Secondary Outcome: CO-confirmed Continuous Abstinence From Week 9 Through Week 24 (Overall)
Description: as for outcome 20
Time Frame: Week 9 through Week 24
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 2037 | 2034 | 2038 | 2035
percentage of participants | 21.8 | 16.2 | 15.7 | 9.4
Statistical Analysis 1: Comparison: Varenicline 1.0 mg BID vs Placebo; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.74, 95% CI 2-sided [2.28 to 3.30]
Statistical Analysis 2: Comparison: Bupropion 150 mg BID vs Placebo; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.56 to 2.29]
Statistical Analysis 3: Comparison: NRT Patch vs Placebo; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.49 to 2.19]

23. Secondary Outcome: 7-Day Point Prevalence of Abstinence, Non-psychiatric History Cohort
Description: A responder to this endpoint requires the answer "no" to both questions 3 and 6 on the nicotine use inventory at that specific visit.
  NUI Question 3 (Baseline through Week 24): Has the subject smoked any cigarettes (even a puff) in the last 7 days? NUI Question 6 (Baseline through Week 12): Has the subject used any other nicotine containing products in the last 7 days? NUI Question 6 (Week 13 through Week 24): Has the subject used any other tobacco products in the last 7 days?
Time Frame: 24 Weeks
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 1005 | 1001 | 1013 | 1009
percentage of participants
  Week 1 | 1.7 | 1.0 | 1.2 | 1.5
  Week 2 | 20.9 | 21.3 | 15.5 | 11.4
  Week 3 | 30.0 | 26.6 | 22.1 | 13.6
  Week 4 | 34.3 | 27.7 | 25.9 | 14.5
  Week 5 | 38.4 | 29.8 | 27.8 | 14.9
  Week 6 | 41.0 | 31.4 | 30.4 | 15.9
  Week 7 | 44.4 | 35.2 | 35.1 | 19.2
  Week 8 | 42.3 | 31.0 | 31.4 | 16.7
  Week 9 | 47.1 | 34.9 | 34.8 | 19.0
  Week 10 | 42.4 | 31.0 | 31.1 | 16.9
  Week 11 | 46.6 | 34.1 | 34.9 | 20.8
  Week 12 | 44.4 | 30.5 | 30.4 | 17.8
  Week 13 | 41.1 | 30.7 | 29.9 | 17.2
  Week 14 | 44.5 | 33.5 | 32.0 | 20.4
  Week 15 | 43.8 | 33.2 | 32.4 | 21.3
  Week 16 | 37.2 | 28.5 | 28.1 | 18.2
  Week 17 | 40.7 | 31.9 | 31.4 | 20.1
  Week 18 | 40.9 | 31.3 | 31.7 | 20.8
  Week 19 | 39.9 | 31.2 | 31.2 | 20.8
  Week 20 | 35.1 | 27.5 | 26.3 | 18.2
  Week 21 | 38.1 | 30.3 | 29.3 | 20.1
  Week 22 | 38.7 | 29.9 | 29.0 | 20.3
  Week 23 | 37.6 | 30.6 | 28.3 | 20.3
  Week 24 | 33.6 | 26.0 | 27.0 | 17.4

24. Secondary Outcome: 7-Day Point Prevalence of Abstinence, Psychiatric History Cohort
Description: as for outcome 23
Time Frame: 24 Weeks
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 1032 | 1033 | 1025 | 1026
percentage of participants
  Week 1 | 1.0 | 1.2 | 0.7 | 0.5
  Week 2 | 16.8 | 14.6 | 13.0 | 9.2
  Week 3 | 22.7 | 18.1 | 17.9 | 10.7
  Week 4 | 26.6 | 21.3 | 21.1 | 11.8
  Week 5 | 28.5 | 21.8 | 22.4 | 12.4
  Week 6 | 30.8 | 22.7 | 23.3 | 13.4
  Week 7 | 34.8 | 25.4 | 27.5 | 16.6
  Week 8 | 32.7 | 22.1 | 24.6 | 15.0
  Week 9 | 36.2 | 26.0 | 29.4 | 17.2
  Week 10 | 35.1 | 24.3 | 25.0 | 14.0
  Week 11 | 38.6 | 27.4 | 29.4 | 17.2
  Week 12 | 35.0 | 23.9 | 24.9 | 14.2
  Week 13 | 32.7 | 22.6 | 24.0 | 14.8
  Week 14 | 34.7 | 25.0 | 26.8 | 17.8
  Week 15 | 33.4 | 25.3 | 26.0 | 18.3
  Week 16 | 29.1 | 21.9 | 21.8 | 13.9
  Week 17 | 32.3 | 24.0 | 24.8 | 17.4
  Week 18 | 31.7 | 24.5 | 24.7 | 18.2
  Week 19 | 31.6 | 24.7 | 25.1 | 17.6
  Week 20 | 26.6 | 20.4 | 25.1 | 17.6
  Week 21 | 29.7 | 23.2 | 23.7 | 17.5
  Week 22 | 29.1 | 22.9 | 23.6 | 16.5
  Week 23 | 28.5 | 23.5 | 22.2 | 16.4
  Week 24 | 26.1 | 20.4 | 20.1 | 14.0

25. Secondary Outcome: 7-Day Point Prevalence of Abstinence (Overall)
Description: as for outcome 23
Time Frame: 24 Weeks
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline 1.0 mg BID | Bupropion 150 mg BID | NRT Patch | Placebo
Number analyzed (Participants) | 2037 | 2034 | 2038 | 2035
percentage of participants
  Week 1 | 1.3 | 1.1 | 0.9 | 1.0
  Week 2 | 18.8 | 17.9 | 14.2 | 10.3
  Week 3 | 26.3 | 22.3 | 20.0 | 12.1
  Week 4 | 30.4 | 24.4 | 23.5 | 13.1
  Week 5 | 33.4 | 25.7 | 25.1 | 13.6
  Week 6 | 35.8 | 26.9 | 26.8 | 14.6
  Week 7 | 39.5 | 30.2 | 31.3 | 17.9
  Week 8 | 37.4 | 26.5 | 28.0 | 15.9
  Week 9 | 41.6 | 30.4 | 32.1 | 18.1
  Week 10 | 38.7 | 27.6 | 28.0 | 15.5
  Week 11 | 42.5 | 30.7 | 32.1 | 18.8
  Week 12 | 39.6 | 27.1 | 27.6 | 16.0
  Week 13 | 36.8 | 26.5 | 26.9 | 16.0
  Week 14 | 39.5 | 29.2 | 29.4 | 19.1
  Week 15 | 38.5 | 29.2 | 29.2 | 19.8
  Week 16 | 33.1 | 25.1 | 24.9 | 16.1
  Week 17 | 36.4 | 27.9 | 28.1 | 18.8
  Week 18 | 36.2 | 27.8 | 28.2 | 19.5
  Week 19 | 35.7 | 27.9 | 28.1 | 19.2
  Week 20 | 30.8 | 23.9 | 23.7 | 16.3
  Week 21 | 33.9 | 26.7 | 26.5 | 18.8
  Week 22 | 33.8 | 26.4 | 26.3 | 18.4
  Week 23 | 33.0 | 27.0 | 25.3 | 18.3
  Week 24 | 29.8 | 23.2 | 23.6 | 15.7

ADVERSE EVENTS:
Time Frame: From baseline throughout the study period (16 weeks). Treatment emergent is first dose date to last dose date (up to 12 weeks) plus 30 days.
Description: AEs were reported from the time the informed consent was signed throughout the study including 30 days after the last dose of study medication. In addition to the the standard collection of volunteered and observed AEs, neuropsychiatric AEs of interest were solicited using the Neuropsychiatric Adverse Event Interview.
Arm/Group | Varenicline 1.0 mg BID | Bupropion | NRT Patch | Placebo
Serious Adverse Events (participants affected / at risk) | 39/2016 | 48/2006 | 45/2022 | 41/2014
Other Adverse Events (participants affected / at risk) | 1158/2016 | 1033/2006 | 1003/2022 | 884/2014
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline 1.0 mg BID (N=2016) | Bupropion (N=2006) | NRT Patch (N=2022) | Placebo (N=2014)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 4 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 1
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 4 | 2
Hernia (General disorders) | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 1 | 0 | 3
Suicide attempt (Psychiatric disorders) | 0 | 2 | 1 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Female sterilisation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 2
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 2 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0
Thyrotoxic crisis (Endocrine disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 3 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 2 | 0 | 0
Bipolar II disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Borderline personality disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
Emotional disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Knee operation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Therapy change (Surgical and medical procedures) | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Vascular rupture (Vascular disorders) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline 1.0 mg BID (N=2016) | Bupropion (N=2006) | NRT Patch (N=2022) | Placebo (N=2014)
Dry mouth (Gastrointestinal disorders) | 66 | 146 | 59 | 64
Nausea (Gastrointestinal disorders) | 511 | 201 | 199 | 137
Application site pruritus (General disorders) | 22 | 12 | 109 | 16
Fatigue (General disorders) | 124 | 57 | 75 | 83
Nasopharyngitis (Infections and infestations) | 174 | 156 | 126 | 135
Upper respiratory tract infection (Infections and infestations) | 109 | 104 | 97 | 115
Headache (Nervous system disorders) | 245 | 186 | 233 | 199
Abnormal dreams (Psychiatric disorders) | 201 | 131 | 251 | 92
Anxiety (Psychiatric disorders) | 132 | 169 | 137 | 120
Insomnia (Psychiatric disorders) | 189 | 245 | 195 | 139
Irritability (Psychiatric disorders) | 82 | 71 | 108 | 104

LIMITATIONS AND CAVEATS:
After database lock and unblinding, one additional participant in the NRT arm of psychiatric cohort was found who had a primary endpoint event (moderate suicidal ideation) which required hospitalization; this event is not included in any analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study participating sites. Investigator may not disclose previously undisclosed confidential other than study results.